CLINICAL TRIAL: NCT00039468
Title: A Phase II Study Of Thalidomide And CPT-11 (IRINOTECAN) Following Radiotherapy For Glioblastoma Multiforme
Brief Title: Thalidomide and Irinotecan in Treating Patients With Glioblastoma Multiforme Who Have Undergone Radiation Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D0134; DMS-15615 (Other: Dartmouth-Hitchcock Medical Center); NCI-G02-2078 (Other Grant/Funding Number: NCI)
Record Dates: First submitted 2002-06-06; First posted 2003-01-27 (Estimated); Last update posted 2011-10-27 (Estimated); Status verified 2011-10

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; recurrent adult brain tumor; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Brain Neoplasms; Gliosarcoma | interventions — Irinotecan; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: irinotecan hydrochloride — 350 or 700 mg/m2 IV every 3 weeks
  Other Names: CAMPTOSAR
Drug: thalidomide — 400mg/day oral
  Other Names: THALOMID

SUMMARY:
RATIONALE: Thalidomide may stop the growth of glioblastoma multiforme by stopping blood flow to the tumor. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining thalidomide with irinotecan may kill any tumor cells remaining after radiation therapy.

PURPOSE: Phase II trial to study the effectiveness of combining thalidomide with irinotecan in treating patients who have glioblastoma multiforme that has been treated with radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate of patients with glioblastoma multiforme treated with thalidomide and irinotecan after radiotherapy.
* Determine the preliminary efficacy of this regimen in these patients.
* Determine the disease-free survival and overall survival of patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.
* Assess the quality of life of patients treated with this regimen.

OUTLINE: Beginning 2-4 weeks after completion of radiotherapy, patients receive irinotecan IV over 90 minutes on day 1. Patients also receive oral thalidomide daily. Treatment repeats every 21 days for at least 3 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, 1 week after the first course, prior to all subsequent courses, and then after course 6.

Patients are followed for 5 years.

PROJECTED ACCRUAL: A total of 9-24 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed glioblastoma multiforme (GBM)

  * Recurrent disease allowed
* Evaluable disease on contrast-enhanced MRI
* Prior external beam radiotherapy required

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST or ALT no greater than 5 times ULN

Renal:

* Creatinine no greater than 1.5 times ULN OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No significant cardiac disease
* No uncontrolled high blood pressure
* No unstable angina
* No congestive heart failure
* No myocardial infarction within the past 3 months
* No serious cardiac arrhythmias

Gastrointestinal:

* Able to take oral medication
* No gastrointestinal abnormalities
* No requirement for IV alimentation
* No active peptic ulcer disease

Other:

* No active infection
* No serious uncontrolled medical disorder
* No dementia or significantly altered mental status that would preclude study
* No known hypersensitivity to irinotecan or thalidomide
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 forms of effective contraception, including 1 highly effective method, at least 1 month before, during, and for 1 month after study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior thalidomide

Chemotherapy:

* No prior irinotecan
* At least 4 weeks since other prior chemotherapy (and demonstrated evidence of disease progression or relapse)

Endocrine therapy:

* Concurrent corticosteroids allowed if on a stable or decreasing dose for at least 1 week prior to study
* No concurrent hormonal therapy for GBM

Radiotherapy:

* See Disease Characteristics
* No concurrent radiotherapy for GBM

Surgery:

* No prior surgical procedures affecting absorption

Other:

* No other concurrent anticancer investigational agents for GBM
* No concurrent cytochrome P450 inhibitors, including the following:

  * Nefazodone
  * Fluvoxamine
  * Fluoxetine
  * Sertraline
  * Paroxetine
  * Venlafaxine
  * Ketoconazole
  * Itraconazole
  * Fluconazole
  * Cimetadine
  * Clarithromycin
  * Diltiazem
  * Erythromycin
  * Protease inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2002-03; Primary Completion 2007-09 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Response | 2 years
  To evaluate the response rate and hence preliminary efficacy of Irinotecan and Thalidomide following radiotherapy in the treatment of newly diagnosed or relapsed glioblastoma multiforme.

SECONDARY OUTCOMES:
Toxicity / QOL / Survival | 2 years
  To evaluate 1) toxicity 2) quality of life 3) disease free survival and 4) overall survival of patients treated with this combination.

CONTACTS AND LOCATIONS:
Overall Officials: Camilo E. Fadul, MD, Study Chair — Norris Cotton Cancer Center
Locations (2):
- United States (2):
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University, Columbus, Ohio

REFERENCES:
- [Result] Fadul CE, Kingman LS, Meyer LP, Cole BF, Eskey CJ, Rhodes CH, Roberts DW, Newton HB, Pipas JM. A phase II study of thalidomide and irinotecan for treatment of glioblastoma multiforme. J Neurooncol. 2008 Nov;90(2):229-35. doi: 10.1007/s11060-008-9655-9. Epub 2008 Jul 26. PMID 18661102